CLINICAL TRIAL: NCT06593314
Title: Identifying Undiagnosed HFpEF Among Patients With Type 2 Diabetes Using Ultromics AI HFpEF Algorithm
Brief Title: Using Ultromics EchoGo HFpEF Algorithm to Identify and Treat High Heart Failure Risk in Patients With Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2024-0209
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Diabetes
Keywords: Subclinical Heart Failure; Electronic Alerts; Diabetes
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Patients with high risk of heart failure (see inclusion/exclusion) as detected by the Ultromics EchoGo algorithm will be included. Each patient will be randomized for their provider to get either a standard message or an Echo-Go message.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EHR Alert Group (Experimental): Provider will receive a computer-based alert notifying them that the patient has subclinical HFpEF as determined by the Ultromics EchoGo algorithm and associated guideline recommendations for the management of these patients. The alert will include guideline-based and standard-of-care recommendations for the use of SGLT-2 inhibitors and/or GLP-1 RA (if obesity is present). The purpose of the alert is to inform the providers about the risk of heart failure and provide them guidance regarding the guideline-recommended standard of care. The providers can choose to provide care as deemed fit based on the information provided
  Interventions: Behavioral: Message with EchoGo
- Standard Message Group (Active Comparator): We will provide a standard message to the provider detailing guideline-recommended medications for type 2 diabetes. This will not contain information about the Ultromics EchoGo algorithm. The providers can choose to provide care as deemed fit based on the information provided
  Interventions: Behavioral: Standard Message

INTERVENTIONS:
Behavioral: Message with EchoGo — This alert will inform the provider that the patient has subclinical HFpEF
  Other Names: EchoGo Message
  Arms: EHR Alert Group
Behavioral: Standard Message — This alert will inform the provider of guideline directed treatment options for patients with diabetes to prevent heart failure.
  Arms: Standard Message Group

SUMMARY:
A pragmatic electronic health record (EHR) based randomized controlled trial to evaluate the utility of providing Ultromics EchoGo analysis results and recommendations for HF risk prevention therapies using an EHR embedded clinical decision support tool.

DETAILED DESCRIPTION:
Historic echocardiograms will be analyzed using the Ultromics EchoGo algorithm. For patients that have a positive EchoGO result i.e. HFpEF detected, the provider will get an clinical decision support alert flagging high risk of HFpEF based on randomized assignment.

Experimental: Alert Group Provider will receive a computer-based provider-to-provider message notifying the provider that the patient has subclinical HFpEF as determined by the Ultromics EchoGo algorithm and associated guideline recommendations for the management of these patients. The alert will include guideline-based and standard-of-care recommendations for the use of SGLT-2 inhibitors, non-steroidal MRA, or GLP-1 RA (if obesity is present). The purpose of the alert is to inform the providers about the risk of heart failure and provide them guidance regarding the guideline-recommended standard of care. The providers can choose to provide care as deemed fit based on the information provided. The investigators will assess the practice patterns of providers in response to the EHR-based alert over the study period (3, and 6-month follow-up). The investigators will also assess the downstream hospitalization events for HF within 12 months of the initial alert.

Control arm: Standard Message Providers in the control group will receive a standard message that will recommend either SGLT2i, GLP-1RA, and/or ns-MRA for treatment of diabetes and for prevention of heart failure. This group will not receive any information about the presence of subclinical heart failure detected by the EchoGo algorithm. The investigators will monitor the practice pattern in this group as well over the study period.

Follow Up. Adherence to SGLT-2i and GLP-1 RA medications will be assessed by evaluating the electronic health record and documenting if the patient had a follow-up with a healthcare provider at 3 and 6 months and medication listed in the active prescription medication list.

Sample Size: The investigators plan to enroll 800 anticipated patients using a parallel design with 1:1 allocation and a binary primary endpoint (SGLT2i use). Using a two-sample test for difference in proportions with the normal (Fleiss) approximation, pooled variance without continuity correction, and assuming a control proportion of 30%, α=0.05 (two-sided), and 80% power, an N=800 (400/arm) provides a minimum detectable absolute increase of ~9.4 percentage points (30.0% to 39.4% in the intervention arm). This corresponds to RR = 1.31(95% CI 1.08, 1.59) and Cohen's h = 0.20.

ELIGIBILITY:
Clinical cohort inclusion exclusion criteria:

Inclusion Criteria:

* Patients with diagnosis of Type 2 diabetes and High WATCH DM score.
* Echocardiogram available in last 6-months.

Exclusion Criteria:

* History of HF
* Not eligible for prescription of new GLP-1RA or SGLT2i or ns-MRA

Corresponding providers to patients identified by the above inclusion exclusion criteria will be included in the clinical trial of the decision support tool.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of prescription of SGLT-2i medication at outpatient clinic visits over 3 months follow-up | 3-month follow-up
  Frequency of prescription of SGLT-2i medication at outpatient clinic visits will be measured as the proportion of new prescription for SGLT2inhibitor divided by the number of alerts triggered.
Frequency of prescription of SGLT-2i medication at outpatient clinic visits over 6 months follow-up | 3-month follow-up
  Frequency of prescription of SGLT-2i medication at outpatient clinic visits will be measured as the proportion of new prescription for GLP1 divided by the number of alerts triggered.

SECONDARY OUTCOMES:
Frequency of prescription of ns-MRA at outpatient clinic visits | 6-months
  Frequency of prescription of ns-MRA at outpatient clinic visits will be measured as the proportion of new prescription for ns-MRA divided by the number of alerts triggered.
Frequency of prescription of GLP-1 RA medication at outpatient clinic visits over | 6 months follow-up
  Frequency of prescription of GLP-1 RA medication at outpatient clinic visits over will be measured as the proportion of new prescription for GLP1 divided by the number of alerts triggered.
Heart Failure hospitalization | 12 months
  Counts of heart failure hospitalization will be recorded form the electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Pandey, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No